CLINICAL TRIAL: NCT00808639
Title: A Phase II Trial of Neoadjuvant Dose-Dense MVAC With Pegfilgrastim Support in Subjects With Muscle-Invasive Urothelial Carcinoma
Brief Title: Dose-Dense MVAC With Pegfilgrastim Support in Subjects With Muscle-Invasive Urothelial Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); Amgen (Industry)
Responsible Party: Principal Investigator, Toni Choueiri, MD, Assistant Professor of Medicine, Harvard Medical School, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-208
Record Dates: First submitted 2008-12-15; First posted 2008-12-16 (Estimated); Results first posted 2014-05-15 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-09

CONDITIONS: Bladder Cancer; Muscle-invasive Bladder Cancer
Keywords: pegfilgrastim; MVAC
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Methotrexate; Doxorubicin; Vinblastine; Cisplatin; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dose Dense MVAC (Experimental): Chemo therapy with methotrexate, vinblastine, Adriamycin, Cisplatin
  Interventions: Drug: Methotrexate; Drug: Doxorubicin; Drug: vinblastine; Drug: cisplatin; Drug: Pegfilgrastim

INTERVENTIONS:
Drug: Methotrexate — intravenously 30mg/m2 over 30 minutes
Drug: Doxorubicin — intravenously 30mg/ms over 15 minutes
Drug: vinblastine — intravenously 3mg/m2 over 30 minutes
Drug: cisplatin — intravenously 70mg/m2 in 1 liter NS with 12.5gm Mannitol over 2 hours after vinblastine completion
Drug: Pegfilgrastim — Given subcutaneously 24 hours after last chemotherapy dose

SUMMARY:
The purpose of this research study is to test the effectiveness of neoadjuvant dose-dense methotrexate, vinblastine, doxorubicin, and cisplatin (ddMVAC) in combination with pegfilgrastim followed by radical surgery in patients with muscle-invasive urothelial carcinoma.

DETAILED DESCRIPTION:
* Participants will be given a study infusion schedule for each treatment cycle. Each treatment cycle lasts three weeks. The infusion of methotrexate will take place on the first day of each cycle. Infusions of vinblastine, doxorubicin and cisplatin will take place on the second day and an injection of pegfilgrastim will be given on the third day.
* During all treatment cycles participants will have a physical exam and will be asked questions about their general health and any problems they might be having and any medications they may be taking.
* Following completion of study treatment, but before surgery, participants will have an assessment of their tumor by CT scan of the chest and and MRI of the abdomen and pelvis.
* Following the participants surgery, we would like to keep track of their medical condition indefinitely, or until this study is officially completed. We would like to do this by calling the participants on the telephone once a year to see how they are doing.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of urothelial cancer. Patients with all histologic subtypes are eligible as long as transitional cell carcinoma is predominant, with the exception of more than a few clusters of small cell carcinoma, which is treated with different chemotherapy and thus are ineligible
* Patients with primary tumors arising in the bladder or urethra are eligible if they have clinical T2-T4a disease
* Patients with primary tumors arising in the ureter or renal pelvis are eligible if they have either grade 3 tumors, or radiographic abnormality large enough to be recognized as an abnormal mass by CT/imaging
* Evaluation by a urologist and be deemed to be acceptable surgical candidates within 3 months of registration
* Adequate physiologic reserves as outlined in the protocol
* Clinical or pathologic N1 lymph node involvement (involvement of a single lymph node < 2cm in greatest dimension) are eligible. Patients with N2-3 or M1 disease are ineligible
* Determination of LV function with an EF > 50%
* Women of child-bearing potential must have a negative pregnancy test
* Patients of child-bearing or father-bearing potential must agree to use an acceptable form of birth control while on the study
* Patients with prior malignancy are eligible provided that the expected outcome from the prior cancer is such that this will not interfere in the delivery of this therapy, or the assessment of response in the cystectomy specimen
* 18 years of age or older

Exclusion Criteria:

* Current, recent (within 3 weeks), or planned participation with other experimental anti-cancer medications as part of clinical trials
* Prior treatment with doxorubicin
* Prior systemic cytoreductive chemotherapy for bladder cancer
* Blood pressure of > 160/100 mmHg. Patients whose blood pressure can be controlled with oral medication are eligible
* NYHA Grade II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 6 months prior to study enrollment
* History of stroke or transient ischemic attack within 6 months prior to study enrollment
* Clinically significant peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Known history of central nervous system or brain metastases
* Major surgical procedure, significant traumatic injury within 21 days prior to Day 1, or anticipation of need for major surgical procedure during the course of the study
* Lactating women
* Patients who are not candidates for surgery, or unwilling to undergo surgery
* Patients with significant fluid collection
* Known hypersensitivity to any component of cisplatin, methotrexate, vinblastine, doxorubicin or pegfilgrastim

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-12; Primary Completion 2013-12 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Toni Choueiri, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choueiri TK, Jacobus S, Bellmunt J, Qu A, Appleman LJ, Tretter C, Bubley GJ, Stack EC, Signoretti S, Walsh M, Steele G, Hirsch M, Sweeney CJ, Taplin ME, Kibel AS, Krajewski KM, Kantoff PW, Ross RW, Rosenberg JE. Neoadjuvant dose-dense methotrexate, vinblastine, doxorubicin, and cisplatin with pegfilgrastim support in muscle-invasive urothelial cancer: pathologic, radiologic, and biomarker correlates. J Clin Oncol. 2014 Jun 20;32(18):1889-94. doi: 10.1200/JCO.2013.52.4785. Epub 2014 May 12. PMID 24821883

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Dense MVAC: Dose-dense methotrexate, vinblastine, doxorubicin, and cisplatin (ddMVAC)
Period: Overall Study
Arm/Group | Dose Dense MVAC
Started | 39
Completed | 38 (One patient went off treatment due to disease progression before surgery.)
Not Completed | 1
Not completed — Disease progression before surgery. | 1

BASELINE CHARACTERISTICS:
Arm/Group | Dose Dense MVAC
Number analyzed (Participants) | 39
Age, Continuous [Median (Full Range); unit: years] | 57 [43 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 39
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Achieving Pathologic Response
Description: Pathological response is defined as down-staging to </=pT1, N0 after chemotherapy with pegfilgrastim support.
Time Frame: After completion of 4 cycles of chemotherapy with pegfilgrastim support (cycle length 2 weeks)
Population: Analysis population consists of all enrolled patients.
Measure: Number (90% Confidence Interval); unit: percentage of pathologic responders
Arm/Group | Dose Dense MVAC
Number analyzed (Participants) | 39
percentage of pathologic responders | 49 [35 to 63]
Statistical Analysis 1: Comparison: Dose Dense MVAC; This study used a Simon's optimal two-stage design. Of 39 eligible patients, if 18 achieved PaR, the treatment would be declared effective. A two-sided 80% CI was estimated considering the two-stage design based on Atkinson and Brown methods; Test type: Superiority or Other; Pathologic response rate = 49, 80% CI 2-sided [38 to 61]

2. Secondary Outcome: Number of Patients Experiencing Febrile Neutropenia
Description: Febrile neutropenia defined per CTCAEv3 as Grade 3 or higher and treatment attribution possibly, probably or definitely-related.
Time Frame: After completion of 4 cycles of chemotherapy with pegfilgrastim support (cycle length 2 weeks)
Measure: Number (90% Confidence Interval); unit: participants
Arm/Group | Dose Dense MVAC
Number analyzed (Participants) | 39
participants | 0 [0 to 0]

3. Secondary Outcome: Number of Patients Experiencing Surgery-related Toxicity
Description: Surgery-related toxicity defined per CTCAEv3 as Grade 2 or higher and treatment attribution possibly, probably or definitely-related.
Time Frame: Surgery + 30 days
Population: Number of patients who underwent cystectomy.
Measure: Number (90% Confidence Interval); unit: participants
Arm/Group | Dose Dense MVAC
Number analyzed (Participants) | 38
participants | 4 [4 to 22]

ADVERSE EVENTS:
Time Frame: Reported adverse events include events starting on or after day 0 through 30 days post treatment.
Description: Toxicities are reported by toxicity type and maximum grade (consolidates the reports of a given type of toxicity for a patient over time) for attributions possibly, probably and definitely related to treatment only. Patients with reports of multiple toxicities of different types are reported multiple times under the relevant toxicity categories.
Arm/Group | Dose Dense MVAC
Serious Adverse Events (participants affected / at risk) | 4/39
Other Adverse Events (participants affected / at risk) | 32/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Dense MVAC (N=39)
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 1
Infection w/ gr3-4 neut, urinary tract (Infections and infestations) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Dense MVAC (N=39)
Tinnitus (Ear and labyrinth disorders) | 1
Opportunistic infection lymphopenia>=gr1 (Infections and infestations) | 1
Phlebitis (Vascular disorders) | 2
Hemoglobin (Blood and lymphatic system disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 3
Chelitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 9
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 3
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 4
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 9
Nausea (Gastrointestinal disorders) | 15
Vomiting (Gastrointestinal disorders) | 4
GI-other (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 27
Edema limb (General disorders) | 1
Pain-other (General disorders) | 1
Infection Gr0-2 neut, mucosa (Infections and infestations) | 1
Infection Gr0-2 neut, oral cavity (Infections and infestations) | 1
Leukocytes (Investigations) | 1
Weight loss (Investigations) | 2
Coagulation-other (Investigations) | 1
ALT, SGPT (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 8
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 1
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 1
Muscle, pain (Musculoskeletal and connective tissue disorders) | 1
Taste disturbance (Nervous system disorders) | 7
Dizziness (Nervous system disorders) | 3
Neuropathy CN I smell (Nervous system disorders) | 1
Neuropathy-sensory (Nervous system disorders) | 1
Head/headache (Nervous system disorders) | 5
Urinary frequency/urgency (Renal and urinary disorders) | 1
Muco/stomatitis (symptom) trachea (Respiratory, thoracic and mediastinal disorders) | 1
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3
Edema, larynx (Respiratory, thoracic and mediastinal disorders) | 1
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes